CLINICAL TRIAL: NCT03605095
Title: Non-invasive Imaging of Human Gingival Microcirculation: Effect of Nitric Oxide
Brief Title: Evidence of Spreading Vasodilation in Human Gingiva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Vag Janos, Principal Investigator, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 5/2018
Record Dates: First submitted 2018-07-11; First posted 2018-07-30 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Nitric Oxide; Vasodilation; Oral Soft Tissue Conditions
Keywords: spreading vasodilation; gingival microcirculation
MeSH Terms: conditions — Aneurysm | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8 mg/ml nitroglycerin (Active Comparator): Higher concentration of NO donor (Nitromint) vs dilution
  Interventions: Drug: nitroglycerin
- 1 mg/ml nitroglycerin (Active Comparator): Lower concentration of NO donor (Nitropohl) vs physiological saline
  Interventions: Drug: nitroglycerin

INTERVENTIONS:
Drug: nitroglycerin — Vasodilatator solution is dropped on the gingiva.

SUMMARY:
The aim of this study is to observe the mechanism of spreading vasodilatation on human healthy gingiva. Nitric-oxide donor solutions in lower and higher concentration are used to trigger the vasoactivity.

DETAILED DESCRIPTION:
Spatial regulation of gingival microcirculation has not been revealed yet. Although this could be an important mechanism to protect gingiva as it is exposed to mechanical, chemical, thermal etc. irritation during whole life. It is especially important during flap surgery. Laser Speckle Contrast Imaging (LSCI) is novel non-invasive method with high spatio-temporal resolution, therefore it allows us to study remote effect of local vasodilation such as spreading vasodilation in human gingiva.

The vasodilatator nitric-oxide (NO) donor will be used to trigger remote effect on gingiva. NO donor solutions will be applied in 1 mg/ml and 8 mg/ml nitroglycerin concentrations. Solution will be dropped on the gingiva at tooth 12 in a fabricated leakage proof well attached to 2mm above the marginal gingiva. The change on blood flow will be monitor at the test well with surrounding gingival area spanning 3 tooth and at the contralateral side by LSCI.

ELIGIBILITY:
Inclusion Criteria:

* general health
* minimum 5 mm keratinized gingiva at upper front teeth

Exclusion Criteria:

* pregnancy and breast-feeding
* medication (except contraceptives)
* smoking
* periodontitis
* caries
* insufficient marginal integrity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Blood flow change after application of NO agonist | 30 min
  The change in blood flow will be measured after locally applied nitroglycerin at the site fo application and at the remote sites

SECONDARY OUTCOMES:
Comparsion of the change in blood flow between genders | 30min
  The maximal blood flow changed assessed in primary outcome will be split into two groups based on gender. The change will be compared between males and females.
Correlation between the change in blood flow and gingival thickness | 30min
  The biotpye will be assessed by measurement of gingival thickness by an ultrasonic devices. The correlation between thickness and maximal vasodilation will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Janos Vag, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided